CLINICAL TRIAL: NCT06722365
Title: Characterization of Fetal Lung With Quantitative Ultrasound
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0634; Protocol Version 1/24/25 (Other: UW Madison); A532860 (Other: UW Madison)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Complication; Fetal Lung Imaging
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- 36 Weeks Pregnant
  Interventions: Device: Backscatter Quantitative Ultrasound

INTERVENTIONS:
Device: Backscatter Quantitative Ultrasound — The intervention consists of a regular abdominal ultrasound scan for fetal evaluation. The difference with a regular scan is that the scanner used to image the fetus provides access to raw/unprocessed ultrasound echo data that can be extracted from the scanner and processed offline (after acquisition) to extract compute backscatter quantitative ultrasound (bQUS) features. Thus, data acquisition does not represent a significant departure from conventional fetal imaging protocols. Other than the time needed to acquire the images, the participant will not perceive any difference from a regular fetal ultrasound scan.
  Other Names: Ultrasound; bQUS

SUMMARY:
The purpose of the study is to show if it's possible to use a special kind of ultrasound called backscatter quantitative ultrasound (bQUS) to check on a baby's lungs when the mother is 36 weeks pregnant. 12 participants will be on study for a single 30 minute ultrasound between 32 and 36 weeks of pregnancy.

DETAILED DESCRIPTION:
Primary Objective:

* Demonstrate the feasibility of performing bQUS analysis on ultrasound echo signals acquired of the fetal lung acquired with clinical ultrasound scanners during third -trimester ultrasound scans

Secondary Objectives:

* Design and implement a protocol to acquire non-processed (raw) echo signals from a commercial ultrasound scanner necessary to perform bQUS at the UPH-Meriter Center for Perinatal Care (CPC).
* Quantify the populational variance of quantitative features extracted from bQUS applied to ultrasound data collected from third trimester ultrasound scans of the fetal lung.

The study will be divided into two phases: (i) feasibility phase and (2) hypothesis-testing phase recruitment phase. Phase 1 will provide evidence of the technical viability of data acquisition at UPH-Meriter CPC and will involve 5 participants. Technical challenges will be discussed with the research team and the supporting vendor (GE) to decide whether the technique is viable to move forward. In case the decision is favorable, recruitment will continue to complete 12 subjects to estimate the populational variance of the quantitative features. If the decision is not favorable due to technical complications, the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females ages 18 to 45 years old with singleton pregnancy, live fetus, gestational age between 32.1 and 36.7 weeks, not in labor, scheduled for routine ultrasound growth evaluation.
* Gestational age determined by the date of the last menses, and confirmed by measurement of the crown-rump-length on transabdominal ultrasound.

Exclusion Criteria:

* Subjects unable to consent.
* Active Labor
* Fetal malformations of the lungs
* Prescription of corticosteroids prior to ultrasound evaluation
* Pre-gestation or gestational diabetes mellitus
* Low English proficiency, needing an interpreter

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant females ages 18 to 45 years old with singleton pregnancy, live fetus, gestational age between 32.1 and 36.7 weeks, not in labor, scheduled for routine ultrasound growth evaluation
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Enrolled as a Proxy for the Feasibility of bQUS to collect technically viable data | data collected over a single study visit (up to 30 minutes)
  Phase 1 will provide evidence of the technical viability of data acquisition at the UPH-Meriter CPC and will involve 5 participants. Technical challenges will be discussed with the research team and the supporting vendor (GE) to decide whether the technique is viable to move forward. In case the decision is favorable, recruitment will continue to complete 12 subjects to estimate the populational variance of the quantitative features. If the decision is not favorable due to technical complications, the study will be terminated.

SECONDARY OUTCOMES:
Population Variance in Fetal Lung Microstructure | data collected over a single study visit (up to 30 minutes)
  Populational variance σ^2_Pop: variance of the individual participant median value of a quantitative ultrasound feature q_(M,s) obtained from the N_S participants included in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: J. Igor Iruretagoyena, MD, MS, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- Meriter Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing with external collaborators will be provided through FlyWheel Exchange.
Time Frame: Coded data and the linking files will be stored for 7 years after conclusion of the study. After seven years, linking files and codes will be destroyed, and the de-identified data will be stored indefinitely for potential future research use.
Access Criteria: Permission to access data will be provided within Data Sharing Agreements and only after IRB approval.